CLINICAL TRIAL: NCT05373641
Title: Effect of Repeated Feedback to RNs' Pain Nursing Documentation: A Cluster Randomized Trial
Brief Title: Effect of Repeated Feedback to Registered Nurses Pain Nursing Documentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Collaborators: University of Eastern Finland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 50UL015
Record Dates: First submitted 2022-02-22; First posted 2022-05-13 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2022-11

CONDITIONS: Education; Nurse's Role; Pain
Keywords: RN; Pain nursing; Pain assessment; Pain management; Pain documentation; Audit and feedback; Education; Randomized Controlled Trial; Nursing sensitive quality; Nursing sensitive outcomes
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: Units serve as a statistical units. Number of units 30, number of individual participants 800-1000.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain documentation audit and repeated feedback (Experimental): Pain documentation audit and repeted feedback
  Interventions: Other: Repeated feedback; Other: Pain documentation audit
- Pain documentation audit (Active Comparator): Pain documentation audit
  Interventions: Other: Pain documentation audit

INTERVENTIONS:
Other: Repeated feedback — Repeated feedback monthly based on previous month pain documentation audit results.
  Arms: Pain documentation audit and repeated feedback
Other: Pain documentation audit — Monthly pain documentation audit

SUMMARY:
The aim of the study is to find out how pain nursing documentation audit and educational feedback effect to RN's pain nursing documentation, the average level of pain nursing documentation knowledge of unit RN's, patient satisfaction of pain management and number of pain nursing incident reports. In addition, how background variables are related to the pain nursing documentation.

Research hypothesis:

Pain nursing documentation audit and educational feedback increased RNs' pain nursing documentation and knowledge, patient satisfaction to pain management and effect to number of pain nursing incident reports.

ELIGIBILITY:
Inclusion Criteria:

* Registered nurses (RN) who work at the Kuopio University Hospital in units of which patients potentially require pain management.

Exclusion Criteria:

* Professionals other than RN
* RN who do not use pain management strategies in their work

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-04 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in RNs' pain documentation | Baseline (T0), month 1 (T1), month 2 (T2), month 3 (T3), month 4 (T4), month 5 (T5) month 6 (T6), month 7 (T7), month 8 (T8)
  MEASUREMENT TOOL: Structured audit frame to evaluate pain assessment and management documentation.
  UNIT OF MEASURE:
  Information is collected as follows from EHR
  1. Patient pain documented in the care chart
  2. Patient need for pain management documented
  3. Patient pain management goal documented
  4. Patient pain assessment
  5. Patient pain assessment in the previous 24 hours
  6. Patient pain
  7. Use of pain assessment tool
  8. Non-pharmacological methods
  9. Pharmacological interventions
  10. Intervention (pharmacological or non-pharmacological effect assessment)
  Multiple measurements are aggregated to achieve one declared value as follows:
  First, each evaluated area results in 0 (not fulfilled) or 1 point (fulfilled). Second, the points are summed. Third, the sum is transformed to a 0-100 scale and reported as a single value reflecting pain documentation quality.
Change in RNs' pain knowledge | Baseline (T0), month 3 (T3), month (T7)
  Pain knowledge questionnaire used in three time points

SECONDARY OUTCOMES:
Change in patient satisfaction of pain management | Before intervention (T0), month 3 (T3), month 6 (T6), month 8 (T8)
  Nursing patient feedback questionnaire analyzed at two time points
Change in number of pain nursing incident reports | Before intervention (T0), month 8 (T8)
  Pain nursing incident reports analyzed at two time points

CONTACTS AND LOCATIONS:
Locations (1):
- Kuopio University Hospital, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grommi S, Voutilainen A, Vaajoki A, Kankkunen P. Effects of Repeated Feedback on Pain Documentation: A Cluster Randomized Trial. Pain Manag Nurs. 2025 Jun;26(3):336-343. doi: 10.1016/j.pmn.2024.12.021. Epub 2025 Jan 30. PMID 39890564